CLINICAL TRIAL: NCT00561678
Title: Perioperative Cognitive Function - Dexmedetomidine and Cognitive Reserve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stacie Deiner, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 06-0217; 1R01AG029656-01A1 (NIH)
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Delirium; PD; Postoperative Cognitive Dysfunction; POCD
Keywords: Postoperative Confusion; Postoperative Delirium; PD; Postoperative Cognitive Dysfunction; POCD
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Precedex (Experimental): Precedex (Dexmedetomidine)
  Interventions: Drug: Precedex (Dexmedetomidine)
- Placebo (Placebo Comparator): Placebo - normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Precedex (Dexmedetomidine) — 0.5/ug/kg/hr Dexmedetomidine infusions will begin prior to the surgery (no loading dose), and will be maintained at 0.5 mcg/kg/hour throughout surgery and titrated postoperatively for 2 hours postoperatively.
  Other Names: Dexmedetomidine
  Arms: Precedex
Drug: Placebo — 0.5/ug/kg/hr Placebo infusions will begin prior to the surgery (no loading dose), and will be maintained at 0.5 mcg/kg/hour throughout surgery and titrated postoperatively for 2 hours postoperatively.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Elderly patients who undergo anesthesia and non-cardiac surgery are subject to deterioration of brain function including the development of postoperative delirium (PD) and postoperative cognitive dysfunction (POCD). These disorders cause disability, distress for both patients and their families, are associated with other medical complications and account for significant additional health care costs. We currently use relatively primitive approaches to preventing and treating PD and POCD.

Dexmedetomidine is a drug used for sedation in critically ill patients that provides some pain relief and controls the bodies response to stress. The sedation produced by dexmedetomidine appears more similar to natural sleep than any other drug used for anesthesia and postoperative sedation. Data suggesting that dexmedetomidine can prevent delirium following cardiac surgery and the developing understanding of the causes of PD and POCD suggest that dexmedetomidine will be particularly effective.

DETAILED DESCRIPTION:
Postoperative Delirium or PD and Postoperative Cognitive Dysfunction or POCD are syndromes of central nervous system dysfunction that significantly complicate the recovery of a proportion of elderly patients following surgery.

Delirium is typically a transient syndrome characterized by a de-novo appearance of several pathognomonic behaviors, including disorientation, decreased attention span, sensory misperceptions, a waxing-and-waning type of confusion, and disorganized thinking. PD typically occurs on postoperative days 1 to 3 and is associated with prolonged hospital stays, increased risks for morbidity and mortality and significant health care expenditures.

The neuroendocrine stress response to surgery, including the immediate postoperative period, remains an important potential etiologic factor. In particular, our data suggests that stress in the immediate postoperative period is poorly controlled by all anesthetic techniques and the normal diurnal variation in cortisol is suppressed in subjects who develop POCD.

Dexmedetomidine is a highly selective alpha 2A agonist currently approved for sedation in the ICU. Dexmedetomidine produces analgesia, sympatholysis, and a light sedation characterized by easy arousal. Its action converges on the endogenous substrates for natural sleep to produce their sedative action, an effect that could prove beneficial to elderly postoperative patients.

We hypothesize that treatment with dexmedetomidine will diminish both PD and POCD. The essential proposition is that modulation of perioperative stress can ameliorate perioperative delirium and cognitive dysfunction.

Based on both the concept of cognitive reserve as well as clinical experience, there is concern that patients with preoperative cognitive impairment are particularly vulnerable to POCD. In general, such patients have been excluded from previous studies. This study is unique in that we will assess all participants for mild cognitive impairment prior to surgery. Assessment of the impact of preexisting cognitive impairment is a secondary aim. A broad goal of this interdisciplinary project is to evaluate POCD, which is primarily an anesthesia concept, in the more general context of dementing illness as explored by geriatric psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* 68 and older
* elective major surgery under general anesthesia(major surgery is defined by a planned 2 day hospitalization)
* ASA physical status I-III
* capable and willing to consent
* MMSE > 20 (to exclude dementia)

Exclusion Criteria:

* Cardiac surgery
* Intracranial Surgery
* Emergency Surgery
* Patients with severe visual or auditory disorder/handicaps
* Illiteracy
* Patients with clinically significant Parkinson's Disease
* Patients not expected to be able to complete the 3 and 6 month postoperative tests
* Sick sinus syndrome without pacemaker
* Hypersensitivity to drug or class
* Current 2nd or 3rd degree AV block
* History of clinically significant bradycardia
* Contraindication to the use of an 2A-agonist
* Presence of a major psychiatric condition such as bipolar disorder, major depression, schizophrenia, or dementia
* ASA physical status IV or V

Min Age: 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 404 (Actual)
Dates: Start 2008-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Silverstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (10):
- United States (10):
  - University of Miami Medical Center, Miami, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - The Mayo Clinic, Rochester, Minnesota
  - St. Louis University, St Louis, Missouri
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Deiner S, Luo X, Lin HM, Sessler DI, Saager L, Sieber FE, Lee HB, Sano M; and the Dexlirium Writing Group; Jankowski C, Bergese SD, Candiotti K, Flaherty JH, Arora H, Shander A, Rock P. Intraoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium and Cognitive Dysfunction in Elderly Patients Undergoing Major Elective Noncardiac Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Aug 16;152(8):e171505. doi: 10.1001/jamasurg.2017.1505. Epub 2017 Aug 16. PMID 28593326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was conducted at 10 sites from February 2008 to May 2014. The lead site was The Mount Sinai Hospital in New York City.
Groups:
- Precedex: Precedex (Dexmedetomidine) 0.5/ug/kg/hr
- Placebo: Placebo - normal saline 0.5/ug/kg/hr
Period: Overall Study
Arm/Group | Precedex | Placebo
Started | 197 | 207
Completed | 189 | 201
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 4 | 3
Not completed — surgery cancelled | 1 | 1
Not completed — surgery rescheduled to different site | 2 | 2
Not completed — anesthesia provider refusal | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Precedex | Placebo | Total
Number analyzed (Participants) | 189 | 201 | 390
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74.0 [71.0 to 78.0] | 74.0 [71.0 to 78.0] | 74.0 [71.0 to 78.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 103 | 200
  Male | 92 | 98 | 190
Education [Median (Inter-Quartile Range); unit: years] | 16.0 [12.0 to 18.0] | 15.0 [12.0 to 17.0] | 16.0 [12.0 to 18.0]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 28.1 [24.3 to 31.7] | 27.7 [24.0 to 32.3] | 28.0 [24.1 to 31.9]
Anesthesia Time [Median (Inter-Quartile Range); unit: minutes] | 252.0 [173.0 to 348.0] | 254.0 [191.0 to 339.0] | 253.0 [185.0 to 345.0]
Surgical Time [Median (Inter-Quartile Range); unit: minutes] | 174.0 [119.0 to 233.0] | 180.0 [123.0 to 249.0] | 177.0 [121.0 to 238.0]
Mild Cognitive Impairment (MCI) [Count of Participants; unit: Participants] | 124 | 122 | 246
ASA Status [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) Physical Status classification:
  1. - normal healthy patient
  2. - patients with mild systemic disease
  3. - patients with severe systemic disease
  4. - patients with severe systemic disease that is a constant threat to life
  Participants
    1 or 2 | 73 | 63 | 136
    3 | 108 | 133 | 241
    4 | 8 | 5 | 13
Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 14 | 18 | 32
Hypertension (HTN) [Count of Participants; unit: Participants] | 124 | 116 | 240
Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] | 0 | 1 | 1
Diabetes (DM) [Count of Participants; unit: Participants] | 39 | 40 | 79
Cancer (CA) [Count of Participants; unit: Participants] | 81 | 77 | 158
Surgical Procedure [Count of Participants; unit: Participants]
  Spine | 70 | 77 | 147
  Thoracic | 5 | 6 | 11
  Orthopedic | 54 | 36 | 90
  Urologic | 20 | 29 | 49
  General | 40 | 53 | 93
Dosage of Fentanyl used prior to this study [Median (Inter-Quartile Range); unit: µg/h] — amount of general anesthesia given
  µg/h | 250.0 [150.0 to 350.0] | 250.0 [200.0 to 400.0] | 250.0 [175.0 to 375.0]
Propofol [Median (Inter-Quartile Range); unit: mg/kg] — amount of general anesthesia given
  mg/kg | 170.0 [120.0 to 360.0] | 160.0 [120.0 to 220.0] | 165.0 [120.0 to 300.0]

OUTCOME MEASURES:

1. Primary Outcome: Delirium Battery
Description: Number of Participants with occurrence of Post-Operative Delirium in Post-Anesthesia Care Unit (PACU)
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Precedex | Placebo
Number analyzed (Participants) | 189 | 201
Participants
  Postoperative Delirium | 23 | 23
  PACU Delirium | 6 | 8
  Both | 5 | 4
  None | 155 | 166

2. Secondary Outcome: Neuropsychological Testing
Description: Rate of change of cognitive function - data not collected because secondary analysis which was not performed
Time Frame: at 3 months postoperatively
Arm/Group | Precedex | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Intraoperative Bradycardia
Description: Number of participants with intraoperative bradycardia
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Precedex | Placebo
Number analyzed (Participants) | 189 | 201
Participants
  Requiring treatment | 35 | 20
  Requiring interruption of the drug | 2 | 2
  Resolved spontaneously | 45 | 42
  Did not occur | 107 | 137

4. Secondary Outcome: Intraoperative Hypotension
Description: Number of participants with intraoperative hypotension
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Precedex | Placebo
Number analyzed (Participants) | 189 | 201
Participants
  Requiring Treatment | 81 | 69
  Requiring interruption of the drug | 3 | 5
  Resolved Spontaneously | 18 | 21
  Did not occur | 87 | 106

5. Secondary Outcome: Intraoperative Hypertension
Description: Number of participants with intraoperative hypertension
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Precedex | Placebo
Number analyzed (Participants) | 189 | 201
Participants
  Requiring treatment | 26 | 36
  Requiring interruption of the drug | 0 | 1
  Resolved spontaneoulsy | 17 | 30
  Did not occur | 146 | 134

6. Secondary Outcome: Length of Stay
Description: Length of Stay (LOS) in the hospital
Time Frame: average 4 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Precedex | Placebo
Number analyzed (Participants) | 189 | 201
days | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 6.0]

ADVERSE EVENTS:
Arm/Group | Precedex | Placebo
All-Cause Mortality (participants affected / at risk) | 1/189 | 3/201
Serious Adverse Events (participants affected / at risk) | 12/189 | 9/201
Other Adverse Events (participants affected / at risk) | 0/189 | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Precedex (N=189) | Placebo (N=201)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Unstable Angina (Cardiac disorders) | 1 | 0
New Arrhythmia (Cardiac disorders) | 2 | 4
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Heart Failure (Cardiac disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Penumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Stroke (Vascular disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 2 | 2
Pulmonary Embolus (Vascular disorders) | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0
GI Bleed (Gastrointestinal disorders) | 1 | 1
Other Infection (Infections and infestations) | 10 | 2
Death (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes